CLINICAL TRIAL: NCT04217863
Title: Effects of the Guided Disclosure Protocol on Post-Traumatic Growth: A Randomized Control Trial Designed to Observe Psychophysiological Alterations in Traumatic Stress Subjects
Brief Title: To Observe the Psychophysiological Alterations in Traumatic Stress Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KU-Psychophysiology-5
Record Dates: First submitted 2019-12-24; First posted 2020-01-06 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Traumatic Stress, Post-Traumatic Growth
Keywords: Guided disclosure protocol; Post-traumatic growth; psycho-physiological alterations; Trauma Symptom Checklist; Sadaf Stress Scale
MeSH Terms: interventions — Guanosine Diphosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental intervention (GDP): It includes three writing (Experimental): 1. Participants will be required to describe memories associated with traumatic event in a sequential order, with an objective and detached attitude
  2. They will be asked to describe
     1. Their opinion regarding the traumatic event and emotions perceived during the experience
     2. Its impact on their daily lives, and how it has altered their attitudes toward life.
  3. The actual situation will be focused, while reviving the whole traumatic event experience which aids in exploring the following aspects:
     * Present thoughts and feelings regarding the traumatic experience, and also clarify the differences between the ones felt at the time of traumatic event in comparison to the current feelings.
     * How much they understand and appreciate themselves for successfully dealing with the traumatic event
     * To what extent the traumatic event has modified their vision, attitude, knowledge, and skills, and how it can help in their future;
     * What will be their future reactions to other similar events.
  Interventions: Behavioral: GDP
- The control intervention: (No Intervention): A day prior to each writing session, the researcher will communicate with each study subject via telephone in order to give them a reminder to perform the writing task and to check their understanding regarding the instructions given in the booklet. Details regarding the inability to contact the subject will also be recorded in the patient form.

INTERVENTIONS:
Behavioral: GDP — Guided Disclosure Protocol
  Arms: The experimental intervention (GDP): It includes three writing

SUMMARY:
This Multicenter study is planned to investigate the effectiveness of the guided disclosure protocol for the promotion of post-traumatic growth (PTG), in the traumatic stress subjects and to determine whether PTG is associated with psychophysiological alterations i.e. (C-Reactive Protein, Brain Derived Neurotropic Factor, Interlukin-6, Cortisol, Heart Rate Variability and brain waves). Study subjects meeting eligibility criteria will be randomized into two groups. Guided disclosure protocol (GDP) will be used as intervention vs the control. Blinded treatment will be provided and the subjects will be made to complete study questionnaires (Screening, Traumatic Stress Scale SSS, Trauma Symptom Checklist, Post-traumatic growth Inventory) at baseline and at post-intervention (3-months later).

DETAILED DESCRIPTION:
Study design:

The study will be conducted as multicenter randomized controlled trial. On the basis of eligibility criteria subjects providing consent to participate in the study will be randomized into two groups, experimental group including those who receive the intervention and a control group receiving control intervention. The study outcomes will be monitored in subjects of both groups at different intervals i.e. at baseline and at 3-month follow-up (post-interventional).

Participants Subjects for the present study will be recruited from 5 centers (based in Karachi, Pakistan). The targeted population includes subjects from diverse ethnicity and considered eligible for participation in the study if they indicated in a pre-screening form that they had experienced traumatic event. These subjects will be invited to participate in the study through advertisement on notice board of each center. A written informed consent will be obtained from each study subject after providing detailed information regarding objectives of the study and its duration.

Interventions

The experimental intervention (GDP):

It includes three writing sessions of 20 minutes where the participants will be made to recall the facts regarding the traumatic event first and then the emotions triggered related to the revealed facts will be channelized. The information related to the immediate priority changes due to the revival of the traumatic history and its reflection on current feelings will be collected. Moreover, the learned coping mechanisms will also be inquired and how the traumatic event altered their vision and their personalities and how it helps in coping with future difficulties.

The original instructions will be translated into local language and altered according to the specific traumatic experience.

In the following, a fusion of the tasks concerning each of the three writing sessions is shown.

1. Participants will be required to describe memories associated with traumatic event in a sequential order, with an objective and detached attitude
2. They will be asked to describe

   1. Their opinion regarding the traumatic event and emotions perceived during the experience
   2. Its impact on their daily lives, and how it has altered their attitudes toward life.
3. The actual situation will be focused, while reviving the whole traumatic event experience which aids in exploring the following aspects:

   * Present thoughts and feelings regarding the traumatic experience, and also clarify the differences between the ones felt at the time of traumatic event in comparison to the current feelings.
   * How much they understand and appreciate themselves for successfully dealing with the traumatic event
   * To what extent the traumatic event has modified their vision, attitude, knowledge, and skills, and how it can help in their future;
   * What will be their future reactions to other similar events. For the writing session it is mandatory to maintain standard experimental environment with maximum silence so that the subject can write peacefully without getting disturbed. Two weeks after the initial assessment, the first writing session will be performed followed by two sessions once every 2 weeks.

The control intervention:

In control intervention the subjects will be required to take three 20-minute writing sessions, in which they will be asked to write about their daily events of the past week, the writing must focus on the facts and highlight an objective and detached attitude. It has shown potential improvements after the guided disclosure protocol (GDP). Works through the placebo effect. Same protocol will be followed for these subjects as the one used for GDP.

A day prior to each writing session, in both conditions either experimental or control the researcher will communicate with each study subject via telephone in order to give them a reminder to perform the writing task and to check their understanding regarding the instructions given in the booklet. Details regarding the inability to contact the subject will also be recorded in the patient form.

ELIGIBILITY:
Inclusion Criteria:

1. Must be disease free, there must be no evidence of any metastatic disease
2. Property of written and spoken the English language.
3. Experienced any traumatic event in the last 12 Months

Exclusion Criteria:

1. Subjects who received a structured psychological intervention for at least 6 months during the last 3 years performed by a psychologist or psychiatrist will be excluded.
2. Those with a codified psychiatric disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) who received Psychopharmacological treatment during the last 3 years will also be excluded from the study sample.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Growth (PTG) | 3 Months
  Change in the Post-traumatic Growth Inventory (PTGI) will be observed among the subjects enrolled in the GDP group as compared to the control group.

SECONDARY OUTCOMES:
C- Reactive Protein (CRP) | 3 Months
  Change in the CRP level will be observed among the subjects enrolled in the GDP group as compared to the control group.
Brain-derived neurotrophic factor (BDNF) | 3 Months
  Change in the BDNF level will be observed among the subjects enrolled in the GDP group as compared to the control group.
Interleukin-6 (IL-6) | 3 Months
  Change in the IL-6 level will be observed among the subjects enrolled in the GDP group as compared to the control group.
Glutamate | 3 Months
  Change in the Glutamate level will be observed among the subjects enrolled in the GDP group as compared to the control group.
Cortisol | 3 Months
  Change in the Cortisol level will be observed among the subjects enrolled in the GDP group as compared to the control group.
Alpha waves | 3 Months
  Change in the Brain waves (Alpha waves) will be observed among the subjects enrolled in the GDP group as compared to the control group.
Heart Rate Variability | 3 Months
  Change in the Heart Rate Variability will be observed among the subjects enrolled in the GDP group as compared to the control group.
Beta waves | 3 Months
  Change in the Brain waves (Beta waves) will be observed among the subjects enrolled in the GDP group as compared to the control group.

OTHER OUTCOMES:
Trauma Symptom Checklist 40 (TSC-40) | 3 Months
  Change in the Trauma Symptom Checklist 40 (TSC-40) will be observed among the subjects enrolled in the GDP group as compared to the control group.
Traumatic Stress Scale (Sadaf Stress Scale) | 3 Months
  Change in the Traumatic Stress Scale will be observed among the subjects enrolled in the GDP group as compared to the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Shamoon Noushad, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandubert C, Scali J, Ancelin ML, Carriere I, Dupuy AM, Bagnolini G, Ritchie K, Sebanne M, Martrille L, Baccino E, Hermes A, Attal J, Chaudieu I. Biological and psychological predictors of posttraumatic stress disorder onset and chronicity. A one-year prospective study. Neurobiol Stress. 2016 Feb 4;3:61-67. doi: 10.1016/j.ynstr.2016.02.002. eCollection 2016 Jun. PMID 27981178
- [Background] Kalisch R, Muller MB, Tuscher O. A conceptual framework for the neurobiological study of resilience. Behav Brain Sci. 2015;38:e92. doi: 10.1017/S0140525X1400082X. Epub 2014 Aug 27. PMID 25158686
- [Background] Cai WP, Pan Y, Zhang SM, Wei C, Dong W, Deng GH. Relationship between cognitive emotion regulation, social support, resilience and acute stress responses in Chinese soldiers: Exploring multiple mediation model. Psychiatry Res. 2017 Oct;256:71-78. doi: 10.1016/j.psychres.2017.06.018. Epub 2017 Jun 8. PMID 28624675
- [Background] Liu AN, Wang LL, Li HP, Gong J, Liu XH. Correlation Between Posttraumatic Growth and Posttraumatic Stress Disorder Symptoms Based on Pearson Correlation Coefficient: A Meta-Analysis. J Nerv Ment Dis. 2017 May;205(5):380-389. doi: 10.1097/NMD.0000000000000605. PMID 27875386
- [Background] Linz R, Puhlmann LMC, Apostolakou F, Mantzou E, Papassotiriou I, Chrousos GP, Engert V, Singer T. Acute psychosocial stress increases serum BDNF levels: an antagonistic relation to cortisol but no group differences after mental training. Neuropsychopharmacology. 2019 Sep;44(10):1797-1804. doi: 10.1038/s41386-019-0391-y. Epub 2019 Apr 16. PMID 30991416
- [Background] Alper B, Erdogan B, Erdogan MO, Bozan K, Can M. Associations of Trauma Severity with Mean Platelet Volume and Levels of Systemic Inflammatory Markers (IL1beta, IL6, TNFalpha, and CRP). Mediators Inflamm. 2016;2016:9894716. doi: 10.1155/2016/9894716. Epub 2016 Apr 5. PMID 27127347
- [Background] Smith HE, Jones CJ, Hankins M, Field A, Theadom A, Bowskill R, Horne R, Frew AJ. The effects of expressive writing on lung function, quality of life, medication use, and symptoms in adults with asthma: a randomized controlled trial. Psychosom Med. 2015 May;77(4):429-37. doi: 10.1097/PSY.0000000000000166. PMID 25939030
- [Background] Gidron Y, Duncan E, Lazar A, Biderman A, Tandeter H, Shvartzman P. Effects of guided written disclosure of stressful experiences on clinic visits and symptoms in frequent clinic attenders. Fam Pract. 2002 Apr;19(2):161-6. doi: 10.1093/fampra/19.2.161. PMID 11906981